CLINICAL TRIAL: NCT00304317
Title: Celecoxib in the Management of Acute Renal Colic
Brief Title: Celecoxib (Celebrex) in the Management of Acute Renal Colic
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI is no longer at the University of Minnesota
Sponsor: University of Minnesota (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0405M60562; 3485B
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Ureteral Calculi
Keywords: calculi; ureteral calculi; ureter
MeSH Terms: conditions — Ureteral Calculi; Calculi | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Celecoxib
  Interventions: Drug: celecoxib
- II (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: celecoxib — Take two capsules (400 mg) by mouth immediately, then take one capsule (200 mg) by mouth every 12 hours until gone.
  Other Names: Celebrex
  Arms: I
Other: Placebo — Take two capsules by mouth immediately, then take one capsule by mouth every 12 hours until gone.
  Arms: II

SUMMARY:
The purpose of this trial is to quantify the amount Celebrex, a specific cyclooxygenase-2 (COX-2) inhibitor, when used for the management of acute renal colic for a ureteral stone will:

* reduce pain medication usage
* improve the percentage of spontaneous stone passage
* decrease the time to spontaneous passage, and
* shift the size distribution of stones passed towards larger sizes

DETAILED DESCRIPTION:
The study will be conducted as a prospective, randomized, double-blind controlled clinical trial. One-hundred and fifty-four patients with symptoms of acute renal colic and a ureteral calculus less than 10 mm in largest diameter on flat plain abdominal x-ray (KUB) or non-contrast computer tomography (CT) scan will be randomized in this trial. At the time of presentation with acute renal colic to the Emergency Department, the patient will be recruited for involvement. After informed consent, patients will be provided either 200 mg of Celebrex or a placebo equivalent. They will be instructed to follow the recommended dosing regimen for acute pain, taking two tablets in the emergency room (400 mg), followed by one tablet 12 hours later (200 mg), then one tablet twice a day for 10 days. Patients will be provided a prescription for Vicodin (1-2 tablets of 5/500 every 4-6 hours) to be taken as required for pain. Throughout the study, patients will be asked to strain urine for passage of calculus and note date and time of passage. Patients will also be asked to maintain a daily narcotic diary and complete a daily pain analog scale provided by our institution. Patients will be followed in the Urology Department's Stone Clinic with weekly imaging studies (KUB or CT scan) and renal function tests (serum creatinine) for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ureteral calculus <= 10 mm in largest diameter
* Patient elects conservative management over immediate surgical intervention

Exclusion Criteria:

* Solitary kidney
* Renal insufficiency (creatinine [CR] > 1.8)
* Urinary infection (fever > 101 degrees Fahrenheit, positive urine culture, many bacteria on urinalysis)
* Allergic-type reactions to sulfonamides
* Patients with known hypersensitivity to celecoxib
* Patients who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or nonsteroidal anti-inflammatory agents (NSAIDs)
* Prior history of gastrointestinal (GI) bleed or active gastric ulcer disease
* Pregnancy/nursing
* Moderate-severe hepatic dysfunction (Child-Pugh Classification B or C)
* Concomitant use of drugs that inhibit P450 2C9, drugs metabolized by P450 2D6, ACE inhibitors, furosemide, warfarin (and other anticoagulants, not including low-dose aspirin), fluconazole, or lithium
* Women of child-bearing age unwilling to use effective contraception for the duration of the trial.
* Significant or unstable cardiovascular disease defined as:

  * myocardial infarction or stroke less than 3 months prior to the study randomization
  * planned revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass surgery [CABG]) at the time of study screening
  * angina at rest or uncontrolled angina
  * hospitalization or emergency department visits for cardiac-related illness less than 3 months prior to randomization
  * uncontrolled hypertension (defined as systolic blood pressure [BP] > 140 mmHg and/or diastolic BP > 90 mmHg at the baseline visit)
  * evidence of cardiac electrophysiologic instability including history of uncontrolled complex ventricular arrhythmia, uncontrolled atrial fibrillation or flutter, or uncontrolled supraventricular tachycardias with a ventricular response heart rate of > 100 beats per minute (BPM) at rest. (Subjects whose cardiac electrophysiologic instability is controlled with a pacemaker or implantable cardioverter defibrillator (ICD) are eligible.)
  * symptoms, signs or treatment for congestive heart failure (CHF) or known left ventricular dysfunction with ejection fraction < 40%
  * undergone coronary bypass surgery or any major surgery (cardiac or noncardiac) or trauma within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Decrease in narcotic usage | at 48 hours

SECONDARY OUTCOMES:
Increase in the percentage of spontaneous stone passage | 6 weeks
Shift in the size distribution of stones passed towards larger sizes | 6 weeks
Decrease in the time to spontaneous passage | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Monga, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States